CLINICAL TRIAL: NCT02875028
Title: Vorapaxar in the Human Endotoxemia Model A Randomized, Double-Blind, Crossover Study
Brief Title: Vorapaxar in the Human Endotoxemia Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bernd Jilma, Ao.Univ.Prof.Dr.med, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPS_Vorapaxar_1.1
Record Dates: First submitted 2016-06-27; First posted 2016-08-23 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
Keywords: Coagulations; Platelets; Inflammation; endotoxemia; vorapaxar
MeSH Terms: conditions — Inflammation; Endotoxemia | interventions — vorapaxar; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vorapaxar (Experimental): subjects will be treated with 4x2,5mg vorapaxar in empty lactose-starch capsules
  Interventions: Drug: Vorapaxar; Other: LPS
- Placebo (Placebo Comparator): subjects will be treated with 4 empty lactose-starch capsules
  Interventions: Drug: Placebo; Other: LPS

INTERVENTIONS:
Drug: Vorapaxar — 10mg-20mg vorapaxar to achieve >80% thrombin-receptor activated peptide-6 (TRAP) induced platelet inhibition
  Arms: Vorapaxar
Drug: Placebo
  Other Names: capsules consisting of lactose-starch
  Arms: Placebo
Other: LPS — 2ng/kg Lipopolysaccharide as a bolus infusion
  Other Names: Lipopolysaccharide

SUMMARY:
Vorapaxar is a recently approved protease activated receptor - 1 (PAR-1) inhibitor. Platelet inhibition may also exert positive results on coagulation activation and may beneficially influence the inflammatory response. Since vorapaxar is the first available substance of a new class of platelet inhibitors its effects on the human coagulation system and the inflammatory response will be assessed in the well-established human endotoxemia model.

DETAILED DESCRIPTION:
Vorapaxar is a novel platelet inhibitor inhibiting PAR-1. It is the first available substance of a new class of platelet inhibitors blocking the activation of platelets via thrombin or thrombin receptor activating peptides via PAR-1. As platelets contribute to the coagulation activation, i.e. by providing the surface for the assembly of the Tenase complex, and furthermore to the inflammatory response by releasing their stored granula containing promotors of both, inflammation and coagulation, we want to assess the effects of vorapaxar on these in the human endotoxemia model. Sixteen healthy volunteers will be included in this randomized, double-blind, placebo-controlled, single center, crossover trial with a washout period of 8 weeks. This wash out period was chosen based on the long elimination half-life of vorapaxar and to prevent any carry-over effects. After intake of 10mg vorapaxar (-24h) the degree of platelet inhibition will be assessed by whole bood aggregometry and, in case of insufficient platelet inhibition, subjects may receive another 10mg of vorapaxar. A bolus of 2ng/kg bodyweight lipopolysaccharide (LPS) will be infused and blood sampling will be performed at pre-defined time-points. After the washout-period the respective other treatment will be given to subjects.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age

  * ≥60 kg bodyweight
  * Normal findings in medical history and physical examination unless the investigator considers the abnormality to be clinically irrelevant
  * Normal laboratory values unless the investigator considers abnormalities to be clinically irrelevant
  * Willingness to comply with the trial's safety demands (to refrain from excessive sporting activities two weeks after Vorapaxar intake, i.e. full contact sports, climbing, mountain biking etc.)
  * Ability to understand the purpose and nature of the study, as well as the associated risks No planned surgeries or other medical interventions in the planned study period

Exclusion Criteria:

* Intake of any drugs that may interfere with the trial's endpoints or drugs (i.e. platelet inhibitors, anticoagulants, CYP3A4 inhibitors, NSAIDs, selective serotonin reuptake inhibitors, selective noradrenaline and serotonin reuptake inhibitors)

  * Positive results of HIV or hepatitis virology
  * Acute illness with systemic inflammatory reactions
  * Known allergies, hypersensitivities or intolerances to any of the used substances
  * Acute or recent bleeding episodes, increased risk of bleeding at the discretion of the investigator
  * History of stroke, transient ischemic attacks or intracerebral hemorrhage
  * Known coagulation or platelet disorders
  * Participation in an LPS trial within 6 weeks of the first study day
  * Severe liver or kidney dysfunction
  * Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
A manuscript will be published in a peer-reviewed journal, individual data will not be presented unless directly requested from the PI (anonymized data may be made publicly available)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 healthy volunteers participated in this crossover trial.
Groups:
- Vorapaxar, Then Placebo: Subjects randomized to this group received vorapaxar treatment first (10-20mg) plus 2ng/kg bodyweight lipopolysaccharide (LPS) bolus infusion and after a washout period of at least 8 weeks, the placebo treatment (0.9% sodium chloride infusion) plus 2ng/kg bodyweight LPS bolus infusion.
- Placebo First, Then Vorapaxar: Subjects randomized to this group received the placebo treatment (0.9% sodium chloride infusion) plus 2ng/kg bodyweight LPS bolus infusion first, and after a washout period of at least 8 weeks, vorapaxar treatment (10-20mg) plus a 2ng/kg bodyweight LPS bolus infusion.
Period: First Intervention (24 Hours)
Arm/Group | Vorapaxar, Then Placebo | Placebo First, Then Vorapaxar
Started (One subject did not participate in the second study period, therefore only 15 started vorapaxar) | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Vorapaxar, Then Placebo | Placebo First, Then Vorapaxar
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention (24 Hours)
Arm/Group | Vorapaxar, Then Placebo | Placebo First, Then Vorapaxar
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: subjects will be treated with 4 empty lactose-starch capsules
  Placebo
  LPS: 2ng/kg Lipopolysaccharide as a bolus infusion
- Total: Total of all reporting groups
Arm/Group | Vorapaxar | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [30 to 36] | 27 [22 to 31] | 31 [27 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 8 | 8 | 16
weight [Median (Inter-Quartile Range); unit: kg] | 70 [64 to 84] | 84 [73 to 88] | 77 [67 to 88]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Prothrombin Fragments F1+2
Description: prothrombin fragment F1+2 concentrations, individual maxima were compared between both study periods
Time Frame: Time points for evaluation were: baseline, 0h, 2h, 4h, 6h, 24h
Population: This was a crossover trial, so all subjects were to complete both study periods (vorapaxar and placebo period). The results of those periods were compared with each other. One subject withdrew during the washout period and was excluded from analysis.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Groups:
- Vorapaxar: Intervention: 10(-20)mg vorapaxar and 2ng/kg bodyweight LPS bolus infusion
- Placebo: Intervention: placebo tablet intake (lactose starch) and 2ng/kg bodyweight LPS bolus infusion
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 16
pmol/L | 1315 [835 to 1800] | 2530 [1175 to 3895]
Statistical Analysis 1: Comparison: Vorapaxar vs Placebo; Test type: Superiority; p = 0.029, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Protease Activated Receptor (PAR)-1 Expression on Platelets
Description: Protease Activated Receptor (PAR)-1 expression on platelets was measured by flow cytometric analysis. The change in protease activated receptor (PAR)-1 expression over time was assessed. The ratio of protease activated receptor (PAR)-1 expression from baseline to 4h was the main parameter of interest and is presented here.
  Since the presented data are ratios, the arbitrary unit is "fold". Otherwise flow cytometric data is presented as "hits" during the analysis.
Time Frame: Time points for evaluation were: baseline, 0h, 4h, 24h
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold
Groups:
- Vorapaxar: Intervention: 10(-20mg) vorapaxar and 2ng/kg bodyweight LPS bolus infusion
- Placebo: Intervention: placebo tablets and 2ng/kg bodyweight LPS bolus infusion
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
fold | 0.85 [0.78 to 1.01] | 0.83 [0.77 to 0.89]

3. Secondary Outcome: Thrombin-Antithrombin Complexes
Description: Thrombin-Antithrombin Complexes were quantified using commercially available "ELISA" assays.
  The individual maxima during the study periods were compared.
Time Frame: Time points for evaluation were: baseline, 0h, 2h, 4h, 6h, 24h
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µg/L
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
µg/L | 17.4 [8.06 to 25.1] | 32.3 [13.9 to 55.2]

4. Secondary Outcome: Plasmin-Antiplasmin Complexes
Description: Plasmin-Antiplasmin Complexes were quantified using commercially available "ELISA" assays. Individual maxima during both study periods were compared.
Time Frame: Time points for evaluation were: baseline, 0h, 2h, 4h, 6h, 24h
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µg/L
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
µg/L | 745 [625 to 1227] | 1437 [764 to 1951]

5. Secondary Outcome: E-Selectin
Description: E-Selectin concentrations were quantified using commercially available "ELISA" assays, individual maxima were compared between both study periods
Time Frame: Time points for evaluation were baseline, 2h, 4h, 6h, 24h after LPS administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
ng/mL | 43.5 [39.85 to 89] | 76.5 [48 to 92.5]

6. Secondary Outcome: Von Willebrand Factor
Description: von Willebrand factor concentrations were measured by commercially available "ELISA" assays, individual maxima were compared between both study periods. The result of this assay are % of "normal" (100%) for this specific assay. The unit therefore is %.
Time Frame: Time points for evaluation were baseline, 2h, 4h, 6h, 24h after LPS administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: % of "normal"
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
% of "normal" | 162 [122 to 193] | 234 [151 to 279]

7. Secondary Outcome: P-Selectin
Description: P-Selectin is quantified using commercially available "ELISA" assays, individual maxima were compared between both study periods.
Time Frame: Time points for evaluation were baseline, 2h, 4h, 6h 24h after LPS administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
ng/ml | 30.8 [21.6 to 33.9] | 33.1 [22.4 to 37.9]

8. Secondary Outcome: Interleukin 6
Description: interleukin-6 concentrations were measured by commercially available "ELISA" assays, individual maxima were compared between both study periods
Time Frame: Time points for evaluation were baseline, 2h, 4h, 6h 24h after LPS administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 105 [74 to 193] | 180 [72 to 370]

9. Secondary Outcome: Tumor Necrosis Factor Alpha
Description: tumor necrosis factor alpha concentrations were measured using commercially available "ELISA" assays, individual maxima were compared between both study periods
Time Frame: Time points for evaluation were: baseline, 0h, 2h, 4h, 6h, 24h
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 27 [13 to 70] | 75 [22 to 96]

10. Secondary Outcome: C-reactive Protein
Description: C-reactive protein levels were measured in the certified central laboratory of the General Hospital, 24h values were compared with each other
Time Frame: Time points for evaluation were: baseline, and 24h after LPS administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
mg/dL | 1.53 [1.15 to 2.19] | 2.44 [1.57 to 2.82]

11. Secondary Outcome: Platelet Factor 4
Description: platelet factor 4 concentrations were quantified by "ELISA", individual maxima were compared between both study periods
Time Frame: Time points for evaluation were: baseline, 0h, 2h, 4h, 6h, 24h
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 53310 [36757 to 73273] | 59803 [39446 to 138624]

12. Secondary Outcome: Thrombomodulin
Description: thrombomodulin concentrations were measured by commercially available "ELISA" assays, individual maxima were compared between both study periods
Time Frame: Time points for evaluation were: baseline, 0h, 2h, 4h, 6h, 24h
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 15 | 15
ng/mL | 5.05 [4.46 to 5.77] | 5.29 [4.58 to 5.49]

ADVERSE EVENTS:
Arm/Group | Vorapaxar | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 11/15 | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorapaxar (N=15) | Placebo (N=16)
headache (Nervous system disorders) | 8 (8) | 5 (5)
Dizziness (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (4) | 7 (7)
Myalgia (General disorders) | 2 (2) | 5 (5)
malaise (General disorders) | 2 (2) | 0 (0)
exanthema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes